CLINICAL TRIAL: NCT02771925
Title: Treatment for Alcohol Dependence With Gabapentin: A Double Blind Placebo Controlled Randomized Clinical Trial
Brief Title: Treatment for Alcohol Dependence With Gabapentin
Acronym: TAG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to poor compliance of patients in the study.
Sponsor: Dayanand Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Prof. Sandeep S Sidhu, Professor Department of Gastroenterology, Dayanand Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAG2016
Record Dates: First submitted 2016-04-18; First posted 2016-05-13 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Alcohol Dependence
Keywords: Gabapentin; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Gabapentin; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gabapentin (Experimental): Total subjects 100 (Alcoholic liver disease:Alcoholics with no liver disease= 1:1) each will receive Gabapentin 2g/day divided in two doses for 24 weeks All patient will receive standard of care treatment
  Interventions: Drug: Gabapentin 2g/day divided in two doses for 24 weeks
- Placebo (Placebo Comparator): Total subjects 100 (Alcoholic liver disease: Alcoholics with no liver disease= 1:1)) each will receive Placebo 2g/day divided in two doses for 24 weeks All patient will receive standard of care treatment
  Interventions: Drug: Placebo 2g/day divided in two doses for 24 weeks

INTERVENTIONS:
Drug: Gabapentin 2g/day divided in two doses for 24 weeks — Total subjects 100 (Alcoholic liver disease:Alcoholics with no liver disease= 1:1) each will receive Gabapentin 2000mg/day divided in two doses for 24 weeks.
  All patients will receive standard of care treatment.
  Other Names: Gabapentin
  Arms: gabapentin
Drug: Placebo 2g/day divided in two doses for 24 weeks — Total subjects 100 (Alcoholic liver disease: Alcoholics with no liver disease= 1:1)) each will receive Placebo 2000mg/day divided in two doses for 24 weeks. All patients will receive standard of care treatment. Concurrent with study medication, study clinicians will provide participants with 20 minutes of weekly manual-guided counseling designed to increase motivation, abstinence, and medication compliance.
  Other Names: Starch
  Arms: Placebo

SUMMARY:
Alcohol use disorders are present across medical specialties, with alcohol-related deaths particularly prevalent in the categories of injury, liver cirrhosis, cancer, cardiovascular disease, disorders of the peripheral nerves and of the central nervous system. Alcohol dependence, also referred to as alcohol use disorder, is a chronic, relapsing disorder marked by compulsive alcohol use, an inability to stop drinking despite harmful consequences, and the emergence of a withdrawal syndrome upon cessation of use. Early abstinence is associated with activation of brain stress systems in the extended amygdala. Clinically, protracted abstinence involves symptoms of craving, mood and sleep disturbance, all of which have been identified as risk factors for relapse. Nonetheless, implementation of alcohol-specific medications remains limited across most medical specialties. Medications for treating alcohol dependence primarily have been adjunctive interventions, and only three medications-disulfiram, naltrexone, and acamprosate-are approved for this indication by the United States Food and Drug Administration. Baclofen, an inhibitor of synaptic transmission through spinal reflex arcs via hyper polarization of primary afferent fiber terminals, was originally approved by the Food and Drug Administration in 1977 for use in spasticity associated with neurologic conditions, such as multiple sclerosis and spinal cord lesions. However, due to its pharmacologic properties it has also been investigated for the treatment of alcohol dependence. But in the clinical practice of study physicians, it was observed that most of the patients who were prescribed baclofen for alcohol dependence hit back to alcohol very soon despite being on the drug. Therefore there is a need to search for an alternative drug which could be beneficial for this population of patients. Gabapentin is Food and Drug Administration-approved for the management of epileptic seizures and neuropathic pain. It is believed to act by blocking a specific alpha-2d subunit of the voltage-gated calcium channel at selective presynaptic sites and, as a result, to indirectly modulate Gamma Butyric Acid neurotransmission. Pre-clinical findings indicate that gabapentin normalizes the stress-induced Gamma Butyric Acid activation in the amygdala that is associated with alcohol dependence, and provide an excellent pre-clinical rationale for evaluating gabapentin as a treatment for alcohol dependence. Earlier studies of gabapentin in alcohol dependent subjects, attempting to abstain following withdrawal support the safety and potential efficacy of gabapentin in alcohol dependent patients, but definitive conclusions were limited by either small sample size, methodological, or dosing issues.

DETAILED DESCRIPTION:
The study will be conducted on patients with alcohol dependence admitted or coming to the out patient department. The enrolled subjects will be divided into two groups randomly using computer generated randomization system. Informed consent shall be taken from the patient/nearest relative of the patient for enrollment in the trial.

The study will be conducted in 2 independent groups in the ratio of 1:1 (each consisting of 100 patients). By taking the rate of sustained abstinence of 4.1% in placebo and 17% in 1800 mg arm and an odd's ratio of 4.8, the sample size needed is 88 patients in each arm. at 80% power and an alpha level of 0.05. Investigators will use an uncorrected chi-squared statistic to evaluate this null hypothesis.

Study Methods

Enrollment of patients, assessing eligibility and obtaining informed consent will be carried out by one of the study investigators. Breath Test analyzer will be use for detecting the blood alcohol content from the breath sample.

Study Intervention

The patients will be randomized to either

Arm A, Total subjects 100 (Alcoholic liver disease:Alcoholics with no liver disease= 1:1) each will receive Gabapentin 2000mg/day divided in two doses for 24 weeks.

All patients will receive standard of care treatment.

or

Arm B, Total subjects 100 (Alcoholic liver disease: Alcoholics with no liver disease= 1:1)) each will receive Placebo 2000mg/day divided in two doses for 24 weeks.

All patients will receive standard of care treatment.

Concurrent with study medication, study clinicians will provide participants with 20 minutes of weekly manual-guided counseling designed to increase motivation, abstinence, and medication compliance.

Laboratory tests

Hemogram, biochemical tests including blood glucose, liver function tests, prothrombin time, serum electrolytes, blood urea and serum creatinine will be done at baseline and subsequently at the end of 1 month, 3 months and 6 months.

Alcohol Breath Test

All the participants will undergoing alcohol breath-testing at monthly for 6 months. A breath-test will be considered positive if a participant submits a test greater than 0.01% Blood Alcohol Concentration. If a result greater than 0.01% Blood Alcohol Concentration is returned the test will be re-administered (the second testing) 15 minutes after the initial test. A proforma including the date, time of breath-test, breath-test reading and signature and name of person administering the breath-test will be maintained.

Follow-up

All patients will be followed up to 6 months or until death. The status alive or dead will be assessed by telephoning a family member or by contacting the death registry at the patient's birth place or place of residence.

ELIGIBILITY:
Inclusion Criteria:

1. Age more then 18 years
2. Meet the Diagnostic and Statistical Manual-Fourth Edition (DSM-V) criteria for current alcohol dependence

Exclusion Criteria:

1. Risk for significant withdrawal based on a Clinical Institute Withdrawal Assessment-Alcohol, Revised (CIWA-AR) score >9
2. More than one month of abstinence
3. Dependence on substances other than alcohol
4. A urine drug screen positive for benzodiazepines or opiates
5. Clinically significant medical or psychiatric disorders treatment with medications that could affect study outcomes
6. Treatment mandated by a legal authority

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Rate of no Heavy Episodic Drinking over 6 month. | 6 month
  (Pattern of reduced drinking, described as no heavy episodic drinking. Heavy episodic drinking days are defined by the FDA - National Institute on Alcohol Abuse and Alcoholism (NIAAA) as days when the patient consumes more than four standard drinks (men) or more than three standard drinks (women). Responder analysis will be applied to the rate of Heavy Episodic Drinking.

SECONDARY OUTCOMES:
Alcohol Craving | 6 month
  Drinking urges were assessed by self-report using the Alcohol Craving Questionnaire-Short Form.
Change in Quality of Life | 6 month
  Mood was evaluated by self report with the Beck Depression Inventory II
Change in sleep pattern | 6 month
  Multiple components of sleep disturbance were assessed by self-report using the Pittsburgh Sleep Quality Index
Rate of Hospital Admission due to alcohol abuse/ decompensation of liver disease | 6 month
Change in Gamma-Glutamyl Transferase (GGT) level over the 6 month period | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep S Sidhu, DM, Principal Investigator — Dayanand Medical College and Hospital, Ludhiana, Punjab, India
Locations (1):
- Dyanand Medical College and Hospital, Ludhiana, Punjab, India

REFERENCES:
- [Result] Mason BJ, Quello S, Goodell V, Shadan F, Kyle M, Begovic A. Gabapentin treatment for alcohol dependence: a randomized clinical trial. JAMA Intern Med. 2014 Jan;174(1):70-7. doi: 10.1001/jamainternmed.2013.11950. PMID 24190578
- [Result] Williams SH. Medications for treating alcohol dependence. Am Fam Physician. 2005 Nov 1;72(9):1775-80. PMID 16300039
- [Result] Rehm J, Mathers C, Popova S, Thavorncharoensap M, Teerawattananon Y, Patra J. Global burden of disease and injury and economic cost attributable to alcohol use and alcohol-use disorders. Lancet. 2009 Jun 27;373(9682):2223-33. doi: 10.1016/S0140-6736(09)60746-7. PMID 19560604
- [Result] Mark TL, Kassed CA, Vandivort-Warren R, Levit KR, Kranzler HR. Alcohol and opioid dependence medications: prescription trends, overall and by physician specialty. Drug Alcohol Depend. 2009 Jan 1;99(1-3):345-9. doi: 10.1016/j.drugalcdep.2008.07.018. Epub 2008 Sep 25. PMID 18819759
- [Result] Koob GF. A role for brain stress systems in addiction. Neuron. 2008 Jul 10;59(1):11-34. doi: 10.1016/j.neuron.2008.06.012. PMID 18614026